CLINICAL TRIAL: NCT02933021
Title: Understanding Monoclonal Gammopathy of Unknown Significance (MGUS): A Research Study to Investigate the Functional Consequences of Paraprotein Production in MGUS
Brief Title: Unravel MGUS (Monoclonal Gammopathy of Unknown Significance)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: RxCelerate Ltd (Industry)
Collaborators: RxCelerate Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: HAF 01; 193751 (Other: IRAS (Integrated Research Application System)); 16/EE/0071 (Other: East of England - Cambridge South Research Ethics Committee)
Record Dates: First submitted 2016-09-15; First posted 2016-10-14 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Monoclonal Gammopathy of Unknown Significance
Keywords: MGUS
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Nurse visit for blood sample, questionnaire and phone call
  Interventions: Other: Blood sample taken; Other: Answering a lifestyle questionnaire; Other: Follow-up phone call from researcher (two years after first visit)

INTERVENTIONS:
Other: Blood sample taken
Other: Answering a lifestyle questionnaire
Other: Follow-up phone call from researcher (two years after first visit) — To enquire about status of participants monoclonal gammopathy of unknown significance, and whether there has been progression to multiple myeloma.

SUMMARY:
This is a study to investigate the functional consequences of paraprotein production in MGUS (Monoclonal Gammopathy of Unknown Significance).

DETAILED DESCRIPTION:
Monoclonal gammopathy of unknown significance (MGUS) is a common haematological condition. It is characterised by proliferation of a B lymphocyte clone and it's associated antibody (paraprotein). In most cases there are no clinical symptoms, however, in a small number of individuals there may be an interaction of the paraprotein with a molecule expressed by the body (self antigen). This can have effects on the normal function of this molecule and/or cause disease.

The study aims to investigate the functional consequences of paraprotein production in MGUS.

ELIGIBILITY:
Inclusion Criteria:

Participants must comply with the following criteria in order to be eligible for the study:

* Be aged ≥18 years at the time the informed consent form is signed
* Have a confirmed and documented Monoclonal Gammopathy of Unknown Significance (MGUS) diagnosis
* Read and understood the participant information sheet, and signed an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved informed consent form prior to any study- specific evaluation

Exclusion Criteria:

Participants will be excluded from joining the study if they match any of the criteria below:

* Pre-existing diagnosis of myeloma/lymphoma
* Participation in a therapeutic clinical study within 28 days or (5 half lives, whichever is longer) of enrolment or during this study
* Any other reason the Clinical Investigator (CI) considers the participant should not join the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit patients diagnosed with Monoclonal Gammopathy of Unknown Significance.
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2016-07; Primary Completion 2019-02-28 (Actual); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical assays (i.e. Haematology, biochemistry, immunology, endocrinology): to capture the number of assay phenotypes that are statistically different from normal ranges. | Up to 4 years from study start
  For clinical assays with defined normal ranges, we will capture those results that are significantly outside of normal range. For those with no generally accepted normal ranges, the results will be compared against results from the other individuals.

SECONDARY OUTCOMES:
The number of conversions to multiple myeloma | 2 years after the first visit

CONTACTS AND LOCATIONS:
Overall Officials: Jill Reckless, Principal Investigator — RxCelerate Limited
Locations (9):
- United Kingdom (9):
  - Royal Berkshire Hospital, Reading, Berkshire
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Torbay Hospital, Torquay, Devon
  - Heartlands Hospital, Birmingham, West Midlands
  - St James's Hospital, Leeds, West Yorkshire
  - Guy's and St. Thomas' Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Rotherham Hospital, Rotherham

IPD SHARING:
Plan to Share IPD: No